CLINICAL TRIAL: NCT00219466
Title: A Parallel, Evaluator-Blind, Randomized Clinical Trial to Evaluate the Efficacy and Safety of Two Marketed Topical Skin Protectants Containing Zinc Oxide in Children With Diaper Rash
Brief Title: Clinical Study to Evaluate the Efficacy and Safety of Two Marketed Investigational Products in Children With Diaper Rash
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A2301007
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2011-08

CONDITIONS: Diaper Rash
MeSH Terms: conditions — Diaper Rash

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Other: Zinc Oxide Diaper Rash Ointment
- 2 (Active Comparator)
  Interventions: Other: Aloe Vera/Tocopherol/Zinc Oxide Cream

INTERVENTIONS:
Other: Zinc Oxide Diaper Rash Ointment — Desitin Original at diaper change
  Other Names: Desitin Original, Formula 311-2
  Arms: 1
Other: Aloe Vera/Tocopherol/Zinc Oxide Cream — Desitin Creamy at diaper change
  Other Names: Desitin Creamy, Formula 316-1
  Arms: 2

SUMMARY:
To evaluate whether Desitin; Zinc Oxide Diaper Rash Ointment (Desitin Original) and Desitin Creamy; Zinc Oxide Diaper Rash Ointment (Desitin Creamy) provide relief of the signs and symptoms associated with diaper rash after 12 and 24 hours of product application.

DETAILED DESCRIPTION:
Subjects received applications of the investigational products following a gentle cleansing of the diaper zone at every diaper change and following bathing of the child during a 24 hour period.

Efficacy was assessed during this study through the documentation of the severity of diaper rash. Results of five anatomic areas and overall severity score by the evaluator's assessments, and parent/guardian's assessments all indicated that both products were significantly effective (P<0.05 in relieving diaper dermatitis (rash) after 12 and 24 hours of treatment.

Safety was assessed through the reporting of adverse events during the course of the study. Overall, the reporting of no adverse events under the conditions of the protocol indicate that the investigational products would appear to be safe for their intended use.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female children, 2-36 months of age
* Wear diapers 24 hours per day
* Present to the test facility for enrollment at baseline with diaper rash receiving an "Overall Severity Score" greater than or equal to 1.5 as determined by the trained evaluator
* Parent/guardian signed informed consent
* Parent/guardian willing to use only the test product in the diaper area during the trial
* Parent/guardian willing to ensure that their child continues to wear their usual brand of diapers and will continue to clean their child during diaper changes using their usual products and method with the exception of ointments, lotions, creams or powders during the trial
* Parent/guardian is willing to refrain from changing any other products whose use may have an effect on their child's skin condition during the trial, i.e., laundry detergents, fabric softeners, and products used to bathe the child
* A Fitzpatrick Skin Type of I-IV

Exclusion Criteria:

* Illness within 4 days preceding enrollment
* Currently being toilet trained
* Active dermatological conditions other than diaper rash that may affect trial results
* History of recurrent dermatological conditions other than diaper rash that may affect trial results
* Concomitant use of medications that may affect trial results
* Known sensitivity to ingredients in trial medications
* Known sensitivity, rash or other abnormal skin reaction to topical or systemic medications or cleansing products within one year of trial initiation
* Other severe acute or chronic medical conditions that may increase the risk associated with trial participation or may interfere with the interpretation of results

Ages: 2 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2005-06; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Trained evaluator's assessment of the severity of diaper rash and Parent/guardian's assessment of response to treatment | At baseline and at 12 and 24 hours post-baseline

SECONDARY OUTCOMES:
Adverse Events | during the course of the study

CONTACTS AND LOCATIONS:
Overall Officials: Qing Li, MD PhD, Study Director — JJCPPW
Locations (1):
- JJCPPW Investigational Site, St. Petersburg, Florida, United States